CLINICAL TRIAL: NCT07043530
Title: Effect of a Sleep Hygiene-based Intervention on Sleep Quality and Mental Health in Medical Students: a Comparison Between In-person and Online Learning
Brief Title: Effect of a Sleep Hygiene-based Intervention on Sleep Quality and Mental Health in Medical Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Yucatán (Other)
Responsible Party: Principal Investigator, Andrea Morales-Robles, Ph.D. student, Universidad Autónoma de Yucatán
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fmed-07-25
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sleep Quality; Mental Health; Students, Medical
Keywords: Sleep hygiene; Sleep quality; Mental health; Medical students; Online intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being; Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person intervention (Active Comparator)
  Interventions: Behavioral: In-person sleep hygiene-based intervention
- Online intervention (Experimental)
  Interventions: Behavioral: Online sleep hygiene-based intervention

INTERVENTIONS:
Behavioral: In-person sleep hygiene-based intervention — The in-person sleep hygiene-based intervention will be delivered in 8 sessions by an sleep expert using digital resources, previously designed and expert validated. During the intervention, the following topics will be covered: (1) sleep hygiene generalities, (2) sleep and environment, (3) sleep and technology, (4) sleep and diet, (5) sleep and excercise, (6) sleep and stimulus control, (7) breathing techniques, (8) mindfulness. The sessions will be delivered twice a week with an approximated duration of 45 minutes each, until completed.
  Arms: In-person intervention
Behavioral: Online sleep hygiene-based intervention — The online sleep hygiene-based intervention will be delivered in 8 sessions through a self-paced educational platform; the content will be the same as in the in-person intervention, but tailored for use in digital learning platforms. The suggest completion time for each session will be 45 minutes. Although its self-paced nature, participants are required to complete it within one month, following the same timeline as the face-to-face arm.
  Arms: Online intervention

SUMMARY:
The aim of the study is to investigate whether an online sleep hygiene programm is as effective as a face-to-face programm in improving sleep quality and mental health in medical students.

ELIGIBILITY:
Inclusion Criteria:

* Being a medical student enrolled in the Universidad Autonoma de Yucatan.
* Having poor sleep quality according to the Pittsburgh Sleep Quality Index.
* Having at least one electronic device with Internet access.
* Having time availability.
* Having signed the informed consent.

Exclusion Criteria:

* Being in their year of Internship or Social Service.
* Being pregnant.
* Having children of any age.
* Being under psychological therapy.
* Regulary consuming sleep, depression or anxiety medication.
* Working the night shift.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | 6 months
  This outcome will be measured by means of the Pittsburgh Sleep Quality Index, which is a self-administered 19-item questionnaire regarding perceived sleep quality, sleep latency, sleep duration, sleep efficiency, sleep alterations, sleep medication use and daytime sleepiness. A score under 6 points suggests good sleep quality, while a score greater or equal to 6 point suggests poor sleep quality.
Mental health | 6 months
  This outcome will be measured by means of the Positive Mental Health Scale (PMHS) and Symptom Checklist 90 Revised (SCL-90-R). The PMHS is a self-administered 83-item questionnaire regarding cognitive and emotional well-being, environmental mastery, social abilities, social sensitivity and empathy, physical well-being, self-reflection, psychological discomfort. The minimum score is 83 and the maximum score is 415; a higher score mean higher positive mental health.
  The SCL-90-R is a self-administered 90-item questionnaire regarding somatization, obssesive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism. Each dimension is independently scored, with a higher grade meaning the pressence of psychological disorders in the evaluated dimension.

OTHER OUTCOMES:
Sleep hygiene | 6 months
  This outcome will be evaluated using the Sleep Hygiene Index.

CONTACTS AND LOCATIONS:
Overall Officials: Héctor A Rubio-Zapata, Dr., Study Director — Universidad Autónoma de Yucatán; Damaris F Estrella-Castillo, Dr., Study Director — Universidad Autónoma de Yucatán
Locations (1):
- Universidad Autónoma de Yucatán, Mérida, Mexico

IPD SHARING:
Plan to Share IPD: Undecided